CLINICAL TRIAL: NCT02881710
Title: Variation IGFBP7 Markers and TIMP2 Induced by Injection of Contrast Iodized Drug at the Intensive Care Patient
Acronym: ContraCHECK
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC14_0241
Record Dates: First submitted 2016-08-24; First posted 2016-08-29 (Estimated); Last update posted 2021-09-21 (Actual); Status verified 2016-08

CONDITIONS: Emergency
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: contrast product used to assess biomarkers variations

SUMMARY:
Multicenter, prospective, uncontrolled study to evaluate variations in urinary concentrations of TIMP-2 and PCI IGFBP7 induced injection during a CT scan in intensive care patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or more,
* Hospitalized in intensive care,
* Holders of a urinary catheter
* Patient receiving a first CT with intravenous injection of PCI during their ICU stay.
* Patient agreeing to participate in the research protocol

Exclusion Criteria:

* Anuria
* Need to retain urine, whatever the reason (eg measurement of 24-hour proteinuria).
* Urine unanalyzable whatever reason (eg urinary washing with double current probe, injection is saline to measure bladder pressure.).
* Patient subjected to renal replacement
* Patient already included in the study for a previous injection of PCI in intensive care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Medical and surgical intensive care adult patients undergoing CT with PCI intravenous injection.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-04-09 (Actual); Primary Completion 2016-03-27 (Actual); Study Completion 2016-03-27 (Actual)

PRIMARY OUTCOMES:
significant increase in urinary concentrations of TIMP-2 and IGFBP7 defined as an increase of NephroCheck® test of more than 0.2 [ng / mL] 2/1000) after PCI injection | follow up: 5 days after injection

IPD SHARING:
Plan to Share IPD: No